CLINICAL TRIAL: NCT02436837
Title: Applicability of Kinect Sensor® in the Rehabilitation of Balance in the Elderly
Acronym: AKS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Juiz de Fora (Other)
Responsible Party: Principal Investigator, Fernando de Sá Silva, PhD, Federal University of Juiz de Fora
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFJFGV0001
Record Dates: First submitted 2015-04-30; First posted 2015-05-07 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Balance; Elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- young (Active Comparator): 20 to 30 years old individuals used as a comparator for elderly group
  Interventions: Other: sessions with virtual reality
- elderly (Experimental): target of treatment to improve the balance.
  Interventions: Other: sessions with virtual reality

INTERVENTIONS:
Other: sessions with virtual reality — sessions with virtual reality to improve the balance

SUMMARY:
Background:

Taking into consideration the ongoing inversion of the population pyramid and the limitations and medical conditions, which predispose to episodes of falling among elderly people, the implementation of exercises and physical treatments capable of promoting postural balance in the group studied is made necessary.

Objectives:

Assess the influence of the electronic platform Kinect Sensor® (KS) as a tool in the treatment of postural balance in elderly individuals. Method: The study included 10 elderly (60 to 70 years old) and 10 young (20 to 30 years old) individuals. Treatment protocol composed of five weeks with sessions performed twice a week with application of KS. Initial and final evaluation included static and dynamic balance instruments: Berg Balance scale and Timed up and Go and Romberg Tandem tests.

DETAILED DESCRIPTION:
Sample Each volunteer has agreed to participate of this research after signing a informed consent. The present work has been approved by the Ethics Committee of Research of the School of Medical and Health Sciences of Juiz de Fora, SUPREMA University, Juiz de Fora, Brazil, under the statement 0015/12.

Each subject filled adequately an anamnesis questionnaire composed of items which referred to the inclusion and exclusion criteria. Those considered incapable of performing activities involving maintenance of balance or belonging to the health risk group were excluded. Health risk was defined by criteria such as, cardiopathies, uncontrolled hypertension, auditory and visual impairment, neurological disturbances and severe muscle-skeletal conditions. Besides those factors, scores inferior to 45 points in the Berg Balance Scale also resulted in exclusion.

In order to collect data, 26 individuals from the Hospital and Maternity Ward Therezinha de Jesus (School of Medical and Health Sciences of Juiz de Fora, SUPREMA University, Juiz de Fora, Brazil) were evaluated. Among them, six have been excluded for distinct reasons, such as, abandoning the proposed sessions or presenting risk factors inserted in the exclusion criteria of the study. The experimental group was composed by 10 subjects (eight females) with mean age of 64.5 years old and the control group had other 10 participants (five females) with mean age 23 years.

The sampled individuals were subject to a sequence of tests specifically devised for static and dynamic balance, which could be used as a comparison parameter for postural balance among the individuals. The tests applied were: a) Timed Up and Go test (TUG); b) Romberg Tandem test; c) Berg Balance scale.

Protocol Treatment protocol consisted of 10 sessions with maximal length of 6 minutes for performing activities using the KS. The interval between the evaluations was of five weeks and the sessions took place twice times a week, according to the participant availability. Before the first session and one day preceding the last, the individuals were evaluated in what concerns static and dynamic balance. Arterial pressure (AP) measurement and stretching activity were performed prior to the KS session. Afterwards, AP was again measured.

Berg Balance Scale Berg Balance scale was the main instrument in the assessment of the postural balance, which was also used as exclusion criterion. It is used in the clinical practice, mainly for the elderly population or neurologic disturbed patients, who have been referred to rehabilitation. The test is constituted of 14 ordinary static and dynamic balance tasks, which are related to quotidian life activities, such as getting up, transfer oneself, standing up, reaching for an object and turning. Each task generates a score between zero and four points, so that the total may be of 56 points. Points are subtracted from the total of a task, if the subject needs aid or external support device to accomplish the particular task. According to Berg et al., patient scoring less or equal to 45 are at high risk of falling during ambulation, what justify the exclusion of volunteers to whom was attributed an inferior score aforementioned.

Timed Up and Go Test In order to perform the Timed Up and Go test (TUG), the subject would rise from a chair, walk three meters and return to the chair. The speed of task execution was established by the participant, with no stimulation by use of verbal commands. The time of execution was measured on the initial evaluation and one day past the tenth session.

Romberg TandemTest According to the protocol established by the Romberg Tandem test, the participants remained with the eyes closed in orthostatic position, with the calcaneus bone of the non-dominant foot placed ahead of the toes of the dominant foot, until the loose balance or reach 60 seconds, maximal time.

Arterial Pressure Arterial pressure (AP) was measured before and after each session. Individuals presenting hypertension stage 3 (≥ 180 systolic and ≥ 110 diastolic), which poses a threat to their practicing of physical activity, were withdrawn of the treatment.

Stretching After AP measurement, all subjects were instructed to perform muscular stretching exercises. The activities were performed in an active and assisted fashion, bilaterally, such as lateral cervical flexion, anterior and posterior inclination of the cervical column, orthostatic torso flexion, torso lateral inclination and rotation on the transverse plane. With the upper limbs, the motions proposed were flexion of shoulder and elbow, horizontal adduction of shoulders and flexion and extension of fingers and wrists. The participants also performed global exercises, cross walks, touching the knees with the hands alternately.

Kinect Sensor All the individuals, including the ones placed in the control group, were instructed on the execution of the activities and accompanied through verbal commands. They were positioned in front of the KS with the highest level of Stack em Up mode (available under the title Yourshape: Fitness Evolved®), and should keep static position with upper limbs raised, simulating sustain a platform. Colored boxes fall upon the simulated platform and must be deposited with the lateral inclination of the torso towards left or right, according to visual stimulus from the television, where virtual apertures are opened on alternate sides at the bottom of the screen. Eventually, fiery boxes fall, and it is necessary to raise the inferior limb of the side where the box is falling towards the platform in order to extinguish the fire, thus flexing knee and pelvic region at 90º.

Statistic Analysis D'agostino & Pearson test was applied to verify the normality of the data. The mean analysis was done by paired Student's t-test for parametric data and Wilcoxon test for non-parametric for the data of each group; unpaired Student's t-test was performed for parametric data and Mann Whitney test for non-parametric data between the evaluated groups.

ELIGIBILITY:
Inclusion Criteria:

* individuals have to be elderly (60 to 70 years old) or young (20 to 30 years old).

Exclusion Criteria:

* anamnesis questionnaire: cardiopathies, uncontrolled hypertension, auditory and visual impairment, neurological disturbances and severe muscle-skeletal conditions.
* cores inferior to 45 points in the Berg Balance Scale also resulted in exclusion.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
anamnesis questionnaire for physical health condition | one day
  Those considered incapable of performing activities involving maintenance of balance or belonging to the health risk group were excluded. Health risk was defined by criteria such as, cardiopathies, uncontrolled hypertension, auditory and visual impairment, neurological disturbances and severe muscle-skeletal conditions.
Berg Balance Scale for equilibrium condition | one day
  Scores inferior to 45 points in the Berg Balance Scale also resulted in exclusion

SECONDARY OUTCOMES:
Berg Balance Scale for equilibrium condition | five weeks
  Berg Balance scale was the main instrument in the assessment of the postural balance
Timed Up and Go Test for the performance of physical agility | five weeks
  In order to perform the Timed Up and Go test (TUG), the subject would rise from a chair, walk three meters and return to the chair. The speed of task execution was established by the participant, with no stimulation by use of verbal commands. The time of execution was measured on the initial evaluation and one day past the tenth session.
Romberg TandemTest for equilibrium performance | five weeks
  According to the protocol established by the Romberg Tandem test, the participants remained with the eyes closed in orthostatic position, with the calcaneus bone of the non-dominant foot placed ahead of the toes of the dominant foot, until the loose balance or reach 60 seconds, maximal time

CONTACTS AND LOCATIONS:
Overall Officials: Andre GF Oliveira, PhD, Principal Investigator — Federal University of Juiz de Fora
Locations (1):
- Federal University of Juiz de Fora, Juiz de Fora, Brazil

REFERENCES:
- [Background] Berg KO, Wood-Dauphinee SL, Williams JI, Maki B. Measuring balance in the elderly: validation of an instrument. Can J Public Health. 1992 Jul-Aug;83 Suppl 2:S7-11. PMID 1468055
- [Background] Berg KO, Maki BE, Williams JI, Holliday PJ, Wood-Dauphinee SL. Clinical and laboratory measures of postural balance in an elderly population. Arch Phys Med Rehabil. 1992 Nov;73(11):1073-80. PMID 1444775
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Diamantopoulos II, Clifford E, Birchall JP. Short-term learning effects of practice during the performance of the tandem Romberg test. Clin Otolaryngol Allied Sci. 2003 Aug;28(4):308-13. doi: 10.1046/j.1365-2273.2003.00710.x. PMID 12871243
- [Background] Agrawal Y, Carey JP, Hoffman HJ, Sklare DA, Schubert MC. The modified Romberg Balance Test: normative data in U.S. adults. Otol Neurotol. 2011 Oct;32(8):1309-11. doi: 10.1097/MAO.0b013e31822e5bee. PMID 21892121